CLINICAL TRIAL: NCT00443521
Title: Triamcinolone as Adjunctive Treatment to Laser Panretinal Photocoagulation for Proliferative Diabetic Retinopathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 310/05
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Last update posted 2007-03-06 (Estimated); Status verified 2007-03

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetes Mellitus/ complications; Diabetic Retinopathy; Triamcinolone; Laser coagulation; Tomography, optical coherence
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Complications | interventions — Triamcinolone Acetonide; Intravitreal Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Triamcinolone Acetonide 4 mg intravitreal injection
Procedure: Panretinal photocoagulation

SUMMARY:
The purpose of the study is to evaluate intravitreal injection of triamcinolone acetonide after laser panretinal photocoagulation in the treatment of proliferative diabetic retinopathy.

DETAILED DESCRIPTION:
The current gold standard for the treatment of proliferative diabetic retinopathy is panretinal photocoagulation. Therefore this study is designed using both treatments in the same patient: intravitreal triamcinolone plus panretinal photocoagulation in one eye, compared to panretinal photocoagulation alone in the contralateral eye. These patients had their visual acuity measured and complete ophthalmological examination was performed, including macular slit lamp examination, fluorescein angiography and optical coherence tomography.

Patients with symmetric proliferative diabetic retinopathy without high risk characteristics receive laser therapy in both eyes and triamcinolone injections in one eye. For the triamcinolone injections, numbing drops, antibiotic drops, and drops to dilate the pupil, and possibly and anesthetic injection, are put in the eye before the medicine is injected into the vitreous. Patients return for follow-up visits 1 day, 1 and 4 weeks after the injection, and then 3 and 6 months. Patients whose condition does not improve may undergo new evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Type II Diabetes
* symmetric proliferative diabetic retinopathy without high risk characteristics
* Informed consent signed

Exclusion Criteria:

* previous treatment for diabetic retinopathy
* media opacities that may interfere with clinical, photographically or OCT examinations
* inability to understands the implications of the protocol
* Glaucoma or ocular hypertension
* Any other pathology that could cause retinal alterations
* Patients with any other situation that may interfere in study completion based in Investigator´s opinion

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-03; Study Completion 2006-07

PRIMARY OUTCOMES:
Visual acuity (ETDRS)
Optic coherence tomography
Vitreous haemorrhage

SECONDARY OUTCOMES:
Safety and Tolerance of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Otacílio O Maia Júnior, M.D., Principal Investigator — Retina and Vitreous Service, Department of Ophthalmology. Hospital das Clínicas. University of São Paulo School of Medicine, Brazil; Walter Y Takahashi, M.D., Study Director — Retina and Vitreous Service, Department of Ophthalmology. Hospital das Clínicas. University of São Paulo School of Medicine, Brazil
Locations (1):
- Retina and Vitreous Service, Department of Ophthalmology. Hospital das Clínicas. University of São Paulo School of Medicine, São Paulo, São Paulo, Brazil